CLINICAL TRIAL: NCT04212065
Title: Long Acting Subcutaneous Compared to Short Acting Sublingual Buprenorphine Administration in Pregnant and Lactating Women
Brief Title: Long Acting Subcutaneous vs Short Acting Sublingual Buprenorphine in Pregnant and Lactating Women
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: closed due to new safety concerns of subcutaneous buprenorphine in pregnant patients
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Kara M Rood, MD, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019H0354
Record Dates: First submitted 2019-12-19; First posted 2019-12-26 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Opioid Use Disorder
Keywords: Sublocade; Suboxone
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine; Sublocade; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Intervention Model Description: This study is a randomized, non-blinded single center clinical trial conducted at Ohio State University (OSU) Wexner Medical Center of 139 women with diagnosed Opioid Use Disorder. These women will be randomized between 14 and 27 weeks to one of two groups:
  * Sublingual Suboxone® 8mg twice daily
  * Subcutaneous SublocadeTM of 300mg monthly
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sublingual Suboxone (Active Comparator): Women randomized to sublingual dosing will be provided prescription to fill.
  Interventions: Drug: buprenorphine
- Subcutaneous Sublocade (Active Comparator): Women randomized to subcutaneous administration will have drug administered by nurse during routine prenatal care visits.
  Interventions: Drug: buprenorphine

INTERVENTIONS:
Drug: buprenorphine — To improve compliance with medication assisted therapy, decrease relapse and neonatal abstinence syndrome, we propose a randomized control trial of long acting subcutaneous buprenorphine compared to short acting sublingual buprenorphine/naloxone administration in pregnant and lactating women.
  Other Names: Sublocade, Suboxone

SUMMARY:
This is a non-inferiority, open label, randomized trial of women on buprenorphine Medication Assisted Therapy for opioid use disorder in pregnancy.Patients will be randomized to either the long acting monthly subcutaneous SublocadeTM or to short acting sublingual Suboxone®.

DETAILED DESCRIPTION:
Opioid use disorder increased among pregnant women in recent years, despite an overall decrease in the general population in the same time frame. Given the increased use of buprenorphine for opioid use disorder, it has now become the most commonly misused prescription opioid subtype. Untreated opioid use disorder is associated with worse maternal, fetal, and neonatal outcomes. To improve compliance with medication assisted therapy, decrease relapse and neonatal abstinence syndrome, we propose a randomized control trial of long acting subcutaneous buprenorphine compared to short acting sublingual buprenorphine/naloxone administration in pregnant and lactating women.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-41 years
* Women with a viable singleton or twin intrauterine pregnancy between 14 0/7 and 27 6/7 weeks gestation based on the best obstetric estimate by ACOG (The American College of Obstetricians and Gynecologists) criteria, and are not planning to terminate the pregnancy.
* Diagnosis of moderate to severe Opioid Use Disorder (OUD), as defined by DSM-V criteria. Mild OUD is defined as 2-3 of the following present, moderate OUD with 4-5 of the following present, and severe OUD with 6 or more of the following present:

  * Substance is often taken in larger amounts and/or over a longer period than the patient intended.
  * Persistent attempts or one or more unsuccessful efforts made to cut down or control substance use.
  * A great deal of time is spent in activities necessary to obtain the substance, use the substance, or recover from effects.
  * Craving or strong desire or urge to use the substance
  * Recurrent substance use resulting in a failure to fulfill major role obligations at work, school, or home.
  * Continued substance use despite having persistent or recurrent social or interpersonal problem caused or exacerbated by the effects of the substance.
  * Important social, occupational or recreational activities given up or reduced because of substance use.
  * Recurrent substance use in situations in which it is physically hazardous.
  * Substance use is continued despite knowledge of having a persistent or recurrent physical or psychological problem that is likely to have been caused or exacerbated by the substance.

The diagnosis and the diagnostic criteria will be recorded.

* Willing to be randomized to subcutaneous or sublingual buprenorphine and to comply with study procedures, including weekly Medication Check Visits
* Planning to deliver at OSU Wexner Medical Center
* Enrolled in prenatal outpatient addiction treatment at OSU
* Able to understand the study, and having understood, provide written informed consent in English

Exclusion Criteria:

* Known allergy or adverse reaction to buprenorphine
* Abnormal obstetrical ultrasound suspicious for major congenital abnormality
* Known or suspected fetal aneuploidy (by either CVS (Chorionic Villus Sampling), amniocentesis or cell-free DNA)
* Participation in another trial that may influence the primary outcome, without prior approval
* Participation in this trial in a prior pregnancy
* Higher order pregnancy
* Have a physiological dependence on alcohol or sedatives requiring medical detoxification
* Have a psychiatric condition that, in the judgment of the site medical clinician (MC), would make study participation unsafe or which would make treatment compliance difficult. Examples include:

  * Suicidal or homicidal ideation requiring immediate attention
  * Severe, inadequately-treated mental health disorder (e.g., active psychosis, uncontrolled bipolar disorder)
* Have a medical condition that, in the judgment of the study MC, would make study participation unsafe or which would make treatment compliance difficult. Medical conditions that may compromise participant safety or study conduct include, but are not limited to, allergy/sensitivity to study medications and the following based on clinical labs:

  * aspartate aminotransferase (AST) / alanine aminotransferase (ALT) greater than 5X upper limit of normal
  * serum creatinine greater than 1.5X upper limit of normal
  * total bilirubin greater than 1.5X upper limit of normal
* Currently in jail, prison or any inpatient overnight facility as required by court of law or have pending legal action or other situation (e.g., unstable living arrangements) that, in the judgement of the site investigator, could prevent participation in the study or in any study activities;
* Currently receiving methadone or naltrexone for the treatment of OUD;
* Enrolled in or planning to enroll in treatment beyond the level of 3.1 (clinically managed low-intensity residential services) of the American Society of Addiction Medicine criteria
* Enrolled in or planning to enroll in: a) a trial testing medication for managing OUD during pregnancy; b) research testing an intervention for substance use disorder or NAS (Neonatal Abstinence Syndrome) in their infant unless they are willing to provide a release for the research records.

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only pregnant women with opioid use disorder
Enrollment: 0 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Evaluating the compliance with prescribed medication is not inferior in women assigned to SublocadeTM compared with those to Suboxone®. | Through study completion, an average of 1.5 years
  Compliance will be assessed by urine drug screens during pregnancy and postpartum visits that are positive for buprenorphine, with assessment of the number of drug screens which are negative for illicit drugs out of the total collected during the study period, with a minimum of three drug screens collected.

SECONDARY OUTCOMES:
Evaluating concentration of buprenorphine and metabolites in maternal plasma | Enrollment through four weeks postpartum
  o A weekly blood draw will be collected, with evaluation of drug concentrations at approximate trough and peak levels before and after drug administration. The blood draw around the time of delivery will evaluate the association between drug concentration and neonatal opioid withdrawal syndrome outcomes.
Evaluating concentration of buprenorphine and metabolites in cord plasma | Delivery
  Cord blood will be collected and used to estimate fetal exposure to buprenorphine
Evaluating concentration of buprenorphine and metabolites in breast milk | 1-6 months postpartum
  Breast milk will be collected and used to estimate infant exposure to buprenorphine via breast milk

CONTACTS AND LOCATIONS:
Overall Officials: Kara Rood, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center OB/GYN Maternal and Fetal Medicine, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No